CLINICAL TRIAL: NCT03150121
Title: Identification of Novel Biomarkers for Early Detection of Ovarian Cancer in High-risk and Normal-risk Populations Using Uterine Lavage
Brief Title: Biomarkers for Early Detection of Ovarian Cancer Using Uterine Lavage
Acronym: BEDOCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Rabin Medical Center (Other); Meir Medical Center (Other); Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-13-0930-KL-CTIL
Record Dates: First submitted 2017-05-03; First posted 2017-05-12 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Ovarian Cancer; Ovarian Carcinoma; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; Serous Cystadenocarcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Cystadenocarcinoma, Serous | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ovarian cancer patients (Experimental): High grade ovarian/fallopian tube/primary peritoneal carcinoma patients with current active disease, at any stage and histological type, who have not yet undergone debulking surgery.
  Interventions: Procedure: Uterine lavage; Procedure: Blood sample; Device: Uterine lavage catheter
- Non-malignant controls (Active Comparator): Patients with non-malignant gynecological conditions indicating surgical procedure, either salpingo-oophorectomy, hysterectomy or hysteroscopy.
  Interventions: Procedure: Uterine lavage; Procedure: Blood sample; Device: Uterine lavage catheter
- High risk population (Experimental): Healthy women with genetically high risk for developing ovarian cancer, who have not undergone risk reducing procedure.
  Interventions: Procedure: Uterine lavage; Procedure: Blood sample; Device: Uterine lavage catheter

INTERVENTIONS:
Procedure: Uterine lavage — Uterine lavage is performed using an intrauterine insemination catheter or rigid pipelle uterine sampler. The catheter is inserted into the cervical canal. 10mL of saline are infused into the uterine cavity and fallopian tubes and immediately retrieved.
  Other Names: Tubo-uterine lavage
Procedure: Blood sample — 5-10mL of blood will be drawn from participants.
Device: Uterine lavage catheter — Uterine lavage is performed using an intrauterine insemination catheter or rigid pipelle uterine sampler. The catheter is inserted into the cervical canal. 10mL of saline are infused into the uterine cavity and fallopian tubes and immediately retrieved.
  Other Names: Intrauterine insemination catheter

SUMMARY:
Screening programs for high-grade ovarian carcinoma failed to reduce disease-specific mortality, since they do not offer early enough detection of the disease. Most cases of high grade ovarian cancer develop in the fallopian tubes, hence the universal recommendation for high-risk populations (e.g., BRCA1/2 mutation carriers) is to undergo risk-reducing bilateral salpingo-oophorectomy (RRBSO) around the age of 40. The aims of this trial are: (1) to identify novel early-stage disease biomarkers using liquid biopsies obtained through uterine lavage, and (2) to optimize the technique a of uterine lavage and the processing of the samples for ultimate implementation as a routine diagnostic test for high risk populations.

DETAILED DESCRIPTION:
Brief Summary:

Screening programs for high-grade ovarian carcinoma failed to reduce disease-specific mortality, since they do not offer early enough detection of the disease. Most cases of high grade ovarian cancer develop in the fallopian tubes, hence the universal recommendation for high-risk populations (e.g., BRCA1/2 mutation carriers) is to undergo risk-reducing bilateral salpingo-oophorectomy (RRBSO) around the age of 40. The aims of this trial are: (1) to identify novel early-stage disease biomarkers using liquid biopsies obtained through uterine lavage, and (2) to optimize the technique a of uterine lavage and the processing of the samples for ultimate implementation as a routine diagnostic test for high risk populations.

The end point of the study is sensitivity and specificity of a liquid biopsy test based on uterine lavage for detection of ovarian cancer.

The study enrolls two cohorts:

1. Proof-of-principle cohort - patients with either established ovarian cancer or other, non-malignant, gynecological conditions.
2. High risk cohort - healthy women at genetically high-risk for ovarian cancer who have not undergone RRBSO.

Inclusion criteria include age over 18, ability to read, understand and sign informed consent form, and planned surgical procedure with general anesthesia (for the proof-of-principle cohort), or planned regular gynecological examination due to high-risk for developing ovarian cancer (high risk cohort).

Exclusion criteria include pregnancy or current attempts to conceive, any prior condition that precludes washing of the entire fallopian tubes.

Patients will provide signed informed consent and will undergo uterine lavage which will be performed by a surgeon before surgery, after induction of anesthesia (proof-of-principle cohort), or by a gynecologist during gynecological examination in an office setting (high risk cohort). Uterine lavage is performed using an intrauterine insemination catheter or rigid pipelle uterine sampler. The catheter is inserted into the cervical canal. 10mL of saline are infused into the uterine cavity and fallopian tubes and immediately retrieved. 5-10mL of blood is also collected from each participant. Patients who have undergone the procedure without anesthesia are requested to complete a pain and stress score questionnaire. All patients are asked to allow access of their medical records and pathology reports from past, present and future gynecologic surgeries.

The uterine lavage liquid biopsy samples are centrifuged to eliminate cells and cell debris. Supernatants were aliquoted within 6 hours from the procedure. Microvesicles, total RNA and DNA are isolated according to previously published protocols.

The samples of the proof-of-principle cohort will be used to define an optimized set of assays, measuring either protein-based or nucleic acid-based biomarkers.

The samples of the high risk cohort will be used to test the sensitivity and specificity of the previously defined biomarkers, and to evaluate confounding factors that may affect the accuracy of the test, such as menopausal status and breast cancer endocrine therapy. Each participant will be asked to consent to uterine lavage procedure on subsequent follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject must have all gynecological organs, including: vagina, cervix, uterus, fallopian tubes and ovaries.
* For the proof-of-principle cohort:

  * Subject must have been evaluated for a gynecologic condition, for which the treating physician has determined that a surgical intervention is required. The surgical procedure may be either: hysterectomy, surgical hysteroscopy, or salpingo-oophorectomy.
  * The eligible gynecological diagnoses include: high grade ovarian, fallopian tube or primary peritoneal carcinoma, or any non-malignant gynecologic condition.
* For the high risk cohort:

  * Subject must have an increased risk for developing ovarian cancer, as determined by genetic testing for BRCA1 or BRCA2 mutations, or by family history of at least one first degree relative that has been diagnosed with high grade ovarian cancer.

Exclusion Criteria:

* Subject is pregnant or is currently attempting to conceive.
* Subject has undergone resection of the uterus, fallopian tubes or ovaries.
* Subject is unable to read, understand and sign the informed consent form.
* Subject refuses to allow access to medical records or pathology reports.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Relevant only for female participants
Enrollment: 500 (Estimated)
Dates: Start 2014-06-29 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Ability of uterine lavage-based biomarkers to detect early stage ovarian cancer | 7 years
  Sensitivity and specificity of proteomic and genomic biomarkers measured in uterine lavage liquid biopsies. The samples will be analyzed in a blinded fashion. The pathological data of the patients will be reviewed and the sensitivity/specificity of each biomarker will be calculated

SECONDARY OUTCOMES:
Complications rate of uterine lavage procedure in high risk population | 7 years
  Assessment of complications rate based on patient's questionnaire and medical records
Burden of uterine lavage procedure as routine diagnostic test for high risk population | 7 years
  Assessment of cost-effectiveness of uterine lavage-based diagnostic test for high risk population, including direct and indirect costs

CONTACTS AND LOCATIONS:
Overall Officials: Keren Levanon, MD,PhD, Principal Investigator — Sheba Medical Center; Yfat Kadan, MD, Principal Investigator — Meir Medical Center; Ram Eitan, MD, Principal Investigator — Rabin Medical Center
Locations (4):
- Israel (4):
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bahar-Shany K, Barnabas GD, Deutsch L, Deutsch N, Glick-Saar E, Dominissini D, Sapoznik S, Helpman L, Perri T, Blecher A, Katz G, Yagel I, Rosenblatt O, Shai D, Brandt B, Meyer R, Mohr-Sasson A, Volodarsky-Perel A, Zilberman I, Armon S, Jakobson-Setton A, Eitan R, Kadan Y, Beiner M, Josephy D, Brodsky M, Friedman E, Anafi L, Molchanov Y, Korach J, Geiger T, Levanon K. Proteomic signature for detection of high-grade ovarian cancer in germline BRCA mutation carriers. Int J Cancer. 2023 Feb 15;152(4):781-793. doi: 10.1002/ijc.34318. Epub 2022 Oct 23. PMID 36214786